CLINICAL TRIAL: NCT00227734
Title: Capecitabine and Oxaliplatin Alone or in Combination With Cetuximab as First-Line Treatment for Metastatic EGFR-Positive Colorectal Cancer, A Randomized Multicenter Phase II Trial
Brief Title: Capecitabine and Oxaliplatin With or Without Cetuximab in Treating Patients With Metastatic Colorectal Cancer That Cannot Be Removed By Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SAKK 41/04; EU-20525
Record Dates: First submitted 2005-09-26; First posted 2005-09-28 (Estimated); Last update posted 2012-06-05 (Estimated); Status verified 2012-06

CONDITIONS: Colorectal Cancer
Keywords: stage IV colon cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Capecitabine; Oxaliplatin; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Active Comparator): Patients receive oral capecitabine twice daily on days 1-15 and oxaliplatin IV over 2 hours on day 1.
  Interventions: Drug: capecitabine and oxaliplatin
- Arm II (Active Comparator): Patients receive capecitabine and oxaliplatin as in arm I and cetuximab IV over 1-2 hours on days 1 and 8
  Interventions: Drug: capecitabine and oxaliplatin + cetuximab

INTERVENTIONS:
Drug: capecitabine and oxaliplatin + cetuximab — cetuximab
  Arms: Arm II
Drug: capecitabine and oxaliplatin — capecitabine and oxaliplatin without cetuximab
  Arms: Arm I

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as capecitabine and oxaliplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells. Monoclonal antibodies, such as cetuximab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Cetuximab may also stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. It is not yet known whether giving capecitabine and oxaliplatin together with cetuximab is more effective than capecitabine and oxaliplatin in treating colorectal cancer.

PURPOSE: This randomized phase II trial is studying how well giving capecitabine and oxaliplatin together with cetuximab works compared to capecitabine and oxaliplatin in treating patients with metastatic colorectal cancer that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the efficacy of capecitabine and oxaliplatin with vs without cetuximab in patients with epidermal growth factor receptor-positive metastatic unresectable colorectal cancer.
* Compare the objective response (complete and partial response) in patients treated with these regimens.

Secondary

* Compare the safety of these regimens in these patients.
* Compare the clinical benefit (complete response, partial response, or stable disease for at least 18 weeks) in patients treated with these regimens.
* Compare overall survival, time to progression, and time to treatment failure in patients treated with these regimens.

OUTLINE: This is a multicenter, randomized study. Patients are stratified according to performance status (0 vs 1), type of metastases (synchronous vs metachronous), prior adjuvant chemotherapy (yes vs no), and participating center. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral capecitabine twice daily on days 1-15 and oxaliplatin IV over 2 hours on day 1.
* Arm II: Patients receive capecitabine and oxaliplatin as in arm I and cetuximab IV over 1-2 hours on days 1 and 8.

In both arms, courses repeat every 3 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients will be followed every 3 months for 1 year and then every 6 months thereafter.

PROJECTED ACCRUAL: A total of 74 patients (37 per treatment arm) will be accrued for this study within 1.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed metastatic colorectal cancer

  * Unresectable disease
  * Primary tumor or metastases must be epidermal growth factor receptor-positive by immunohistochemistry
* Measurable disease, defined as ≥ 1 unidimensionally measurable lesion ≥ 20 mm by conventional techniques OR ≥ 10 mm by CT scan

  * Measurable lesion must not be in a previously irradiated area
* No prior or current CNS metastases

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* WHO 0-1

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic

* Bilirubin normal

Renal

* Creatinine clearance > 50 ml/min

Cardiovascular

* No New York Heart Association class III or IV congestive heart failure
* No symptomatic coronary artery disease
* No uncontrolled cardiac arrhythmia
* No myocardial infarction within the past 12 months
* No other significant cardiac disease

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception during and for 12 months after study participation
* Negative pregnancy test
* No peripheral neuropathy of any origin > grade 1 (e.g., alcohol or diabetes)
* No nausea, vomiting, or malabsorption syndrome that would preclude ingestion or absorption of oral medication
* No severe reaction attributed to fluoropyrimidine therapy
* No known hypersensitivity to fluorouracil or any other component of the trial drugs
* No known dihydropyrimidine dehydrogenase deficiency
* No other medical condition (e.g., uncontrolled diabetes or active autoimmune disease), geographical situation, or psychiatric disorder that would preclude study compliance
* No other malignancy within the past 5 years except adequately treated carcinoma in situ of the cervix or localized nonmelanoma skin cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior chemotherapy for advanced or metastatic cancer
* At least 6 months since prior adjuvant chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* At least 30 days since prior experimental drugs
* No other concurrent experimental drugs
* No concurrent drugs that are contraindicated for use with the trial drugs
* No other concurrent anticancer therapy
* No concurrent sorivudine or any of its chemically-related analogues (e.g., lamivudine)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2004-06; Primary Completion 2005-10 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Objective response (complete response [CR] and partial response [PR]) measured after completion of study treatment

SECONDARY OUTCOMES:
Clinical benefit (CR, PR, and stable disease [SD]) measured at 18 weeks after randomization
Time to progression
Overall survival
Time to treatment failure measured after completion of study treatment
Adverse drug reactions measured after completion of study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Markus M. Borner, MD, Study Chair — Insel Gruppe AG, University Hospital Bern; Dieter Koeberle, MD, Principal Investigator — Cantonal Hospital of St. Gallen
Locations (18):
- Switzerland (18):
  - Kantonspital Aarau, Aarau
  - Hirslanden Klinik Aarau, Aarau
  - Praxis Dr. Streit, Baden
  - Kantonsspital Baden, Baden
  - Saint Claraspital AG, Basel
  - Universitaetsspital-Basel, Basel
  - Inselspital Bern, Bern
  - Kantonsspital Bruderholz, Bruderholz
  - Spitaeler Chur AG, Chur
  - Hopital Cantonal Universitaire de Geneve, Geneva
  - Kantonsspital, Liestal
  - Ospedale Civico, Lugano
  - Praxis Dr. Beretta, Rheinfelden
  - Kantonsspital - St. Gallen, Sankt Gallen
  - Regionalspital, Thun
  - City Hospital Triemli, Zurich
  - Stadtspital Waid, Zurich
  - UniversitaetsSpital Zuerich, Zurich

REFERENCES:
- [Result] Borner M, Koeberle D, Von Moos R, Saletti P, Rauch D, Hess V, Trojan A, Helbling D, Pestalozzi B, Caspar C, Ruhstaller T, Roth A, Kappeler A, Dietrich D, Lanz D, Mingrone W; Swiss Group for Clinical Cancer Research (SAKK), Bern, Switzerland. Adding cetuximab to capecitabine plus oxaliplatin (XELOX) in first-line treatment of metastatic colorectal cancer: a randomized phase II trial of the Swiss Group for Clinical Cancer Research SAKK. Ann Oncol. 2008 Jul;19(7):1288-1292. doi: 10.1093/annonc/mdn058. Epub 2008 Mar 17. PMID 18349029